CLINICAL TRIAL: NCT01857297
Title: A Phase IV, Single-Centre, Open-label Study to Evaluate the Immunogenicity and Safety of the 2013/2014 Formulation of the Enzira® Vaccine in Two Groups of Healthy Volunteers: 'Adults' (Aged 18 to 59 Years) and 'Older Adults' (Aged 60 Years or Older).
Brief Title: A Study to Assess the Immunogenicity and Safety of CSL's 2013/2014 Formulation of Enzira® Vaccine in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSLCT-ASU-12-82; 2013-000945-37 (EudraCT Number)
Record Dates: First submitted 2013-05-12; First posted 2013-05-20 (Estimated); Results first posted 2014-01-15 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-04

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adults (aged 18 to 59 years) (Experimental): The study vaccine (Enzira® vaccine) is a sterile, thiomersal-free suspension containing 45 mcg total haemagglutinin antigen per 0.5 mL dose (15 mcg each of the three recommended influenza strains for the Northern Hemisphere 2013/2014 influenza season). The vaccine will be administered by intramuscular or deep subcutaneous injection.
  Interventions: Biological: Enzira® vaccine
- Older Adults (aged 60 years or older) (Experimental): The study vaccine (Enzira® vaccine) is a sterile, thiomersal-free suspension containing 45 mcg total haemagglutinin antigen per 0.5 mL dose (15 mcg each of the three recommended influenza strains for the Northern Hemisphere 2013/2014 influenza season). The vaccine will be administered by intramuscular or deep subcutaneous injection.
  Interventions: Biological: Enzira® vaccine

INTERVENTIONS:
Biological: Enzira® vaccine
  Other Names: Afluria® vaccine

SUMMARY:
This is a study to assess the immune (antibody) response and safety of the 2013/2014 formulation of Enzira® vaccine in healthy adult volunteers aged 18 years or older.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 years or older at the time of vaccination.
* Females of child-bearing potential (i.e., ovulating, pre-menopausal, not surgically sterile) must be abstinent or be willing to use a medically accepted contraceptive regimen for the duration of the study. Females of child-bearing potential must return a negative urine pregnancy test result prior to vaccination with the vaccine.

Exclusion Criteria:

* Known hypersensitivity to a previous vaccination with influenza vaccine or allergy to eggs, ovalbumin, chicken protein, neomycin, polymyxin, or any components of the vaccine.
* Clinical signs of an active infection.
* A clinically significant medical condition.
* Vaccination with a seasonal or experimental influenza virus vaccine in the 6 months preceding study entry.
* Females who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Director Vaccines, Study Director — Seqirus
Locations (1):
- Study Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was non-randomized with a parallel assignment comprising of 2 groups of healthy volunteers: adults (aged 18 - 59 years) and older adults (aged 60 years or older).
Pre-assignment Details: None relevant
Groups:
- Adults (18 to 59 Years): Healthy volunteers aged 18 to 59 years received a single 0.5 mL dose of CSL Influenza Vaccine by intramuscular or subcutaneous injection.
- Older Adults (60 Years or Older): Healthy volunteers aged 60 years or older received a single 0.5 mL dose of CSL Influenza Vaccine by intramuscular or subcutaneous injection.
Period: Overall Study
Arm/Group | Adults (18 to 59 Years) | Older Adults (60 Years or Older)
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adults (18 to 59 Years) | Older Adults (60 Years or Older) | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Customized [Mean (Standard Deviation); unit: years]
  Years | 34.5 (11.17) | 69.4 (6.02) | 51.9 (19.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 30 | 70
  Male | 20 | 30 | 50

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Evaluable Participants Achieving Seroconversion or Significant Increase in Antibody Titre.
Description: As per the criteria specified in the CPMP/BWP/214/96 Note for Guidance on Harmonisation of Requirements for Influenza Vaccines. For haemagglutination inhibition (HI), seroconversion (H1N1, H3N2, and B influenza virus strains) is defined as achieving a post-vaccination titre of ≥ 40 for those participants with a pre-vaccination HI titre of < 10. A significant increase (H1N1, H3N2, and B influenza virus strains) is defined as a four-fold or greater increase in HI titre for those participants with a pre-vaccination HI titre of ≥ 10.
Time Frame: Approximately 21 days after vaccination
Population: The Evaluable Population included all participants who were vaccinated with the Influenza Vaccine, provided both pre- and post-vaccination antibody titer results, did not use a prohibited medication as per the protocol, and were not excluded from the analysis according to the elimination criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adults (18 to 59 Years) | Older Adults (60 Years or Older)
Number analyzed (Participants) | 59 | 60
percentage of participants
  H1N1 strain | 72.9 [59.7 to 83.6] | 63.3 [49.9 to 75.4]
  H3N2 strain | 78.0 [65.3 to 87.7] | 55.0 [41.6 to 67.9]
  B strain | 54.2 [40.8 to 67.3] | 30.0 [18.8 to 43.2]

2. Primary Outcome: The Geometric Mean Fold Increase (GMFI) in Antibody Titre After Vaccination.
Description: GMFI (H1N1, H3N2, and B influenza virus strains) is defined as the geometric mean of the fold increases of post-vaccination antibody titre over the pre-vaccination antibody titre.
Time Frame: Approximately 21 days after vaccination
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: fold increase
Arm/Group | Adults (18 to 59 Years) | Older Adults (60 Years or Older)
Number analyzed (Participants) | 59 | 60
fold increase
  H1N1 strain | 12.90 (4.764) | 6.11 (3.675)
  H3N2 strain | 17.85 (5.237) | 5.77 (4.549)
  B strain | 5.30 (3.522) | 2.81 (2.858)

3. Primary Outcome: The Percentage of Evaluable Participants Achieving a HI Titre ≥ 40 or Single Radial Haemolysis (SRH) Area ≥ 25 mm2.
Description: For the H1N1, H3N2 and B influenza virus strains. Note: No SRH data were collected.
Time Frame: Approximately 21 days after vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adults (18 to 59 Years) | Older Adults (60 Years or Older)
Number analyzed (Participants) | 59 | 60
percentage of participants
  H1N1 strain | 98.3 [90.9 to 100] | 95.0 [86.1 to 99.0]
  H3N2 strain | 100 [93.9 to 100] | 98.3 [91.1 to 100]
  B strain | 86.4 [75.0 to 94.0] | 51.7 [38.4 to 64.8]

4. Secondary Outcome: Frequency of Any Solicited Adverse Events (AEs)
Description: The percentage of participants reporting any solicited AEs.
Time Frame: During the 4 days after vaccination (Day 0 plus 3 days)
Population: The Safety Population included all participants who received the Influenza Vaccine and provided follow-up safety data.
Measure: Number; unit: percentage of participants
Arm/Group | Adults (18 to 59 Years) | Older Adults (60 Years or Older)
Number analyzed (Participants) | 60 | 60
percentage of participants
  Any solicited local AE | 61.7 | 13.3
  Induration > 50 mm | 1.7 | 0
  Erythema | 5.0 | 0
  Ecchymosis | 3.3 | 0
  Pain | 58.3 | 13.3
  Any solicited systemic AE | 25 | 10
  Temperature > 38°C for ≥ 24 hours | 0 | 1.7
  Chills | 10 | 6.7
  Malaise | 23.3 | 6.7

5. Secondary Outcome: Frequency of Any Unsolicited AEs
Description: The percentage of participants reporting any unsolicited AEs. Unsolicited AEs include AEs other than those specifically solicited.
Time Frame: After vaccination until the end of the study; approximately 21 days.
Population: The Safety Population included all participants who received the Influenza Vaccine and provided follow-up safety data.
Measure: Number; unit: percentage of participants
Arm/Group | Adults (18 to 59 Years) | Older Adults (60 Years or Older)
Number analyzed (Participants) | 60 | 60
percentage of participants | 46.7 | 36.7

ADVERSE EVENTS:
Time Frame: For solicited AEs: During the 4 days after vaccination (Day 0 plus 3 days); For unsolicited AEs and serious AEs (SAEs): After vaccination until the end of the study (approximately 21 days).
Description: The other AEs presented include solicited and unsolicited AEs. The Safety Population included all participants who received CSL Influenza Vaccine and provided follow-up safety data.
Arm/Group | Adults (18 to 59 Years) | Older Adults (60 Years or Older)
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 40/60 | 16/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults (18 to 59 Years) (N=60) | Older Adults (60 Years or Older) (N=60)
Injection site pain (General disorders) | 35 (35) | 8 (8)
Malaise (General disorders) | 14 (15) | 4 (5)
Chills (General disorders) | 6 (7) | 4 (5)
Headache (Nervous system disorders) | 15 (17) | 6 (6) — unsolicited adverse event
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (1) — unsolicited adverse event
Pyrexia (General disorders) | 4 (4) | 0 (0) — unsolicited adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.